CLINICAL TRIAL: NCT05823896
Title: An Interventional, Double-Blinded, 2-Arm Study to Investigate the Efficacy of Orally Administered Nirmatrelvir/Ritonavir Compared with Placebo/Ritonavir in Non-hospitalized Adult Participants Suffering from Post-COVID
Brief Title: ImPROving Quality of LIFe in the Long COVID Patient
Acronym: PROLIFIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Petter Brodin, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KI-PROLIFIC-2023; 2022-003855-32 (EudraCT Number)
Record Dates: First submitted 2023-04-20; First posted 2023-04-21 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-09

CONDITIONS: Post-COVID-19 Syndrome; Long COVID; Long Covid19; COVID-19; POTS - Postural Orthostatic Tachycardia Syndrome; Post COVID-19 Condition; Post-COVID Syndrome; Post COVID-19 Condition, Unspecified; Postinfectious Inflammation; Postinfectious Disorder
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Postural Orthostatic Tachycardia Syndrome; Post-Infectious Disorders | interventions — nirmatrelvir and ritonavir drug combination; Ritonavir

STUDY DESIGN:
Intervention Model Description: This is a phase II, interventional, randomized, parallel group, double-blind, placebo-controlled, single-center study of nirmatrelvir/ritonavir (300/100 mg) or placebo/ritonavir (100mg), administered orally twice daily for 15 days in non-hospitalized patients with post- COVID conditions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nirmatrelvir/ritonavir (Active Comparator): Oral nirmatrelvir/ritonavir (Paxlovid) 300/100 mg twice daily for 15 days
  Interventions: Drug: Nirmatrelvir/ritonavir
- Placebo/ritonavir (Placebo Comparator): Oral placebo/ritonavir 100 mg twice daily for 15 days
  Interventions: Drug: Placebo/ritonavir

INTERVENTIONS:
Drug: Nirmatrelvir/ritonavir — 300/100 mg tablet twice daily (q12h) administered orally for 15 days
  Other Names: Paxlovid
  Arms: Nirmatrelvir/ritonavir
Drug: Placebo/ritonavir — 100mg tablet twice daily (q12h) administered orally for 15 days
  Other Names: Placebo
  Arms: Placebo/ritonavir

SUMMARY:
The purpose of this study is to investigate the efficacy of orally administered nirmatrelvir/ritonavir compared with placebo/ritonavir to improve quality of life in non-hospitalized adult participants suffering from post-acute COVID-19 syndrome.

DETAILED DESCRIPTION:
At present there is no curative treatment for post-acute COVID-19 syndrome (PACS). Treatment is focused on symptom management and individualized rehabilitation. There is data indicating SARS-CoV-2 viral persistence and chronic immune system activation in PACS. We are proposing an interventional, randomized and placebo-controlled clinical intervention trial of nirmatrelvir/ritonavir (300/100 mg) or placebo/ritonavir (100mg), twice daily for 15 days, in patients suffering from severe PACS and meeting the WHO definition of severe PACS. A total of 180 patients will be enrolled in this study and these will be randomized in a 2:1 ratio to receive either nirmatrelvir/ritonavir or placebo/ritonavir. The study will include deep exploratory systems-level analyses of the immune system in PACS patients, including changes induced by nirmatrelvir/ritonavir (Paxlovid®) treatment. The purpose of this study is to evaluate the efficacy of nirmatrelvir/ritonavir for its potential ability to provide sustained improvement in quality of life, in non-hospitalized patients with post-COVID, a patient group with high unmet medical needs.

Hypothesis: Nirmatrelvir/ritonavir (Paxlovid®) improves health-related quality of life measured using the EQ-5D-5L VAS scale, as compared to placebo/ritonavir, in objective and pre-defined clinical phenotypes: postural orthostatic tachycardia syndrome (POTS), microvascular dysfunction, inappropriate sinus tachycardia, persistent fever, post exertional malaise (PEM), fatigue, brain fog, dyspnea, dysfunctional breathing patterns or inflammatory phenotypes (increased plasma D-dimer, CRP, ESR and ferritin).

ELIGIBILITY:
Inclusion Criteria:

1. The subject has given written consent to participate in the study.
2. ≥18 years of age at the time of the Screening Visit.
3. Post-acute COVID-19 syndrome (PACS) according to the WHO definition.
4. EQ-5D-5L VAS ≤ 50
5. All fertile participants must agree to use a highly effective method of contraception for the duration of the study and 28 days after last intake of the IMP.

Exclusion Criteria:

General exclusion criteria

1. Other non-related conditions with PACS like symptoms.
2. Renal function eGFR eGFRCysC < 60 mL/min/1.73 m2.
3. Not able to comply with the study protocol.
4. Previous Paxlovid treatment.
5. Pregnancy or breastfeeding.
6. Drug-drug interaction with ongoing treatment, including concomitant use of any medications or substances that are strong inducers of CYP3A4 within 28 days prior to first dose of nirmatrelvir/ritonavir and during study treatment.
7. Participants who are planning or considering vaccination (including boosters) through Study Day 45.
8. Active COVID-19 infection as verified by SARS CoV-2 positive antigen test.
9. Self-reported medical conditions, including:

   1. Type 1 or Type 2 diabetes mellitus.
   2. Chronic kidney disease.
   3. Neurodevelopmental disorders (e.g., cerebral palsy, Down's syndrome) or other conditions that confer medical complexity (e.g., genetic or metabolic syndromes and severe congenital anomalies).
   4. Active cancer other than localized skin cancer, including those requiring treatment including palliative treatment), as long as the treatment is not among the prohibited medications that must be administered/continued during the trial period.
   5. Immunosuppressive disease (e.g., bone marrow or organ transplantation or primary immune deficiencies) OR prolonged use of immune-weakening medications:

   i. Has received corticosteroids equivalent to prednisone ≥20 mg daily for at least 14 consecutive days within 30 days prior to study entry.

   ii. Has received treatment with biologics (e.g., infliximab, ustekinumab, etc.), immunomodulators (e.g., methotrexate, 6MP, azathioprine, etc.), or cancer chemotherapy within 90 days prior to study entry.

   iii. HIV infection with CD4+ cell count <200/mm3.
10. History of hospitalization for the medical treatment of acute COVID-19
11. Current need for hospitalization or anticipated need for hospitalization within 48 hours after randomization in the clinical opinion of the site investigator.
12. Prior/Concomitant Therapy:

    1. Current or expected use of any medications or substances that are highly dependent on CYP3A4 for clearance, and for which elevated plasma concentrations may be associated with serious and/or life-threatening events during treatment and for 4 days after the last dose of nirmatrelvir/ritonavir. List of potential interactions provided by Pfizer provided in Appendix A.
    2. Has received or is expected to receive monoclonal antibody treatment, antiviral treatment (e.g., molnupiravir), or convalescent COVID-19 plasma.

    Prior/Concurrent Clinical Study Experience:
13. Is unwilling to abstain from participating in another interventional clinical study with an investigational compound or device, including those for post-COVID-19 therapeutics, through the long-term follow-up visit.
14. Previous administration with any investigational drug or vaccine within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
15. Known prior participation in this trial or other trial involving nirmatrelvir.

    Diagnostic Assessments:
16. Known history of any of the following abnormalities in clinical laboratory tests (within past 6 months of the screening visit):

    * AST or ALT level ≥2.5 X ULN
    * Total bilirubin ≥2 X ULN (≥3 X ULN for Gilbert's syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in quality of life over time | Baseline and day 16
  The effect of oral administration of nirmatrelvir/ritonavir on quality of life measured as change from baseline using the EQ-5D-5L VAS scale.

SECONDARY OUTCOMES:
Change from baseline in quality of life over time | Baseline and days 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on quality of life measured as change from baseline using the EQ-5D-5L VAS scale.
Change from baseline in hemodynamic response over time | Baseline and days 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on hemodynamic response (only patients diagnosed with postural orthostatic tachycardia syndrome, POTS). Change from baseline in delta maximum heart rate during active standing test.
Change from baseline in dysautonomia over time | Baseline and days 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on dysautonomia symptoms. Change from baseline as measured using the Composite Autonomic Symptom Score (Compass31) questionnaire.
Change from baseline in fever in patients with POTS over time | Baseline and days 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on fever (only patients diagnosed with POTS). Change from baseline in POTS-specific symptoms as measured by using the Malmo POTS score, MAPS.
Change from baseline in endothelial function over time | Baseline and day 45
  The effect of oral administration of nirmatrelvir/ritonavir on reactive hyperemia index. Change from baseline in endothelial function measured using the EndoPat® device.
Change from baseline in heart rate over time | Baseline and days 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on 24-h average heart rate. Change from baseline in heart rate using ECG monitoring device.
Change from baseline in fever over time | Baseline and days 16, 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on fever. Change from baseline in body temperature.
Change from baseline in physical capacity over time | Baseline and days 16, 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on physical capacity. Change from baseline as measured by 6-minute walk test.
Change from baseline in handgrip strength over time | Baseline and days 16, 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on handgrip strength. Change from baseline as measured by JAMAR hand dynamometer.
Change from baseline in physical activity over time | Baseline and days 16, 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on physical activity. Change from baseline as measured by accelerometer.
Change from baseline in post-exertional malaise over time | Baseline and day 90
  The effect of oral administration of nirmatrelvir/ritonavir on post-exertional malaise. Change from baseline in total score as measured by the Post-Exertional Malaise (PEM) short form.
Change from baseline in fatigue over time | Baseline and days 16, 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on fatigue. Change from baseline as measured by the fatigue severity scale (FSS) and mental fatigue scale (MFS).
Change from baseline in cognitive dysfunction over time | Baseline and days 16, 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on cognitive dysfunction. Change from baseline over time as measured by the Montreal Cognitive Assessment (MoCA) test.
Change from baseline in dyspnea over time | Baseline and days 16, 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on dyspnea measured as change from baseline in respiratory symptoms using the Chronic obstructive disease assessment (CAT) and Modified Medical Research Council (mMRC) tests.
Change from baseline in plasma biomarkers over time | Baseline and days 16, 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on plasma biomarkers. Change from baseline in the following plasma biomarkers: D-dimer, CRP, ESR, ferritin, NTproBNP and LD.
Change from baseline in dysfunctional breathing patterns over time | Baseline and days 16, 45 and 90
  The effect of oral administration of nirmatrelvir/ritonavir on dysfunctional breathing patterns. Change from baseline in Njimegen questionnaire.

OTHER OUTCOMES:
Change from baseline in relationships between genotypes and immune function over time | At baseline and day 16
  The effect of oral administration of nirmatrelvir/ritonavir on the relationship between genotypes and immune function at the molecular level. Circulating protein levels adjusted for DNA-variants.
Change from baseline in immune cell function over time | At baseline and day 16
  The effect of oral administration of nirmatrelvir/ritonavir on changes in immune cell function as assessed by high-dimensional cytometry.
Change from baseline in persistence of SARS-CoV-2 virus over time | At baseline and day 16
  The effect of oral administration of nirmatrelvir/ritonavir on persistence of SARS-CoV-2 virus as measured by:
  Protein profiling using Olink Explore Inflammation panel. Nucleosome-profiling (using Volition) and circulating spike (using SIMOA™, Quanterix).
  PBMC profiling for scTCR-sequencing (using BD Rhapsody) with assessment of Super-Ag-mediated T-cell activation.
  Immune system signatures associated with disease states using RNA-sequencing of stabilized whole blood (PaxGene).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Runold, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caruso D, Guido G, Zerunian M, Polidori T, Lucertini E, Pucciarelli F, Polici M, Rucci C, Bracci B, Nicolai M, Cremona A, De Dominicis C, Laghi A. Post-Acute Sequelae of COVID-19 Pneumonia: Six-month Chest CT Follow-up. Radiology. 2021 Nov;301(2):E396-E405. doi: 10.1148/radiol.2021210834. Epub 2021 Jul 27. PMID 34313468
- [Background] Han X, Fan Y, Alwalid O, Li N, Jia X, Yuan M, Li Y, Cao Y, Gu J, Wu H, Shi H. Six-month Follow-up Chest CT Findings after Severe COVID-19 Pneumonia. Radiology. 2021 Apr;299(1):E177-E186. doi: 10.1148/radiol.2021203153. Epub 2021 Jan 26. PMID 33497317
- [Background] Ceban F, Ling S, Lui LMW, Lee Y, Gill H, Teopiz KM, Rodrigues NB, Subramaniapillai M, Di Vincenzo JD, Cao B, Lin K, Mansur RB, Ho RC, Rosenblat JD, Miskowiak KW, Vinberg M, Maletic V, McIntyre RS. Fatigue and cognitive impairment in Post-COVID-19 Syndrome: A systematic review and meta-analysis. Brain Behav Immun. 2022 Mar;101:93-135. doi: 10.1016/j.bbi.2021.12.020. Epub 2021 Dec 29. PMID 34973396
- [Background] Goh D, Lim JCT, Fernaindez SB, Joseph CR, Edwards SG, Neo ZW, Lee JN, Caballero SG, Lau MC, Yeong JPS. Case report: Persistence of residual antigen and RNA of the SARS-CoV-2 virus in tissues of two patients with long COVID. Front Immunol. 2022 Sep 5;13:939989. doi: 10.3389/fimmu.2022.939989. eCollection 2022. PMID 36131932
- [Background] Visvabharathy L, Orban ZS, Koralnik IJ. Case report: Treatment of long COVID with a SARS-CoV-2 antiviral and IL-6 blockade in a patient with rheumatoid arthritis and SARS-CoV-2 antigen persistence. Front Med (Lausanne). 2022 Sep 23;9:1003103. doi: 10.3389/fmed.2022.1003103. eCollection 2022. PMID 36213654
- [Background] Hammond J, Leister-Tebbe H, Gardner A, Abreu P, Bao W, Wisemandle W, Baniecki M, Hendrick VM, Damle B, Simon-Campos A, Pypstra R, Rusnak JM; EPIC-HR Investigators. Oral Nirmatrelvir for High-Risk, Nonhospitalized Adults with Covid-19. N Engl J Med. 2022 Apr 14;386(15):1397-1408. doi: 10.1056/NEJMoa2118542. Epub 2022 Feb 16. PMID 35172054
- [Background] Toussi SS, Neutel JM, Navarro J, Preston RA, Shi H, Kavetska O, LaBadie RR, Binks M, Chan PLS, Demers N, Corrigan B, Damle B. Pharmacokinetics of Oral Nirmatrelvir/Ritonavir, a Protease Inhibitor for Treatment of COVID-19, in Subjects With Renal Impairment. Clin Pharmacol Ther. 2022 Oct;112(4):892-900. doi: 10.1002/cpt.2688. Epub 2022 Jul 5. PMID 35712797
- [Background] Sundaram A, Vaughan B, Kost K, Bankole A, Finer L, Singh S, Trussell J. Contraceptive Failure in the United States: Estimates from the 2006-2010 National Survey of Family Growth. Perspect Sex Reprod Health. 2017 Mar;49(1):7-16. doi: 10.1363/psrh.12017. Epub 2017 Feb 28. PMID 28245088
- [Background] Swank Z, Senussi Y, Manickas-Hill Z, Yu XG, Li JZ, Alter G, Walt DR. Persistent Circulating Severe Acute Respiratory Syndrome Coronavirus 2 Spike Is Associated With Post-acute Coronavirus Disease 2019 Sequelae. Clin Infect Dis. 2023 Feb 8;76(3):e487-e490. doi: 10.1093/cid/ciac722. PMID 36052466
- See also: Recommendations related to contraception and pregnancy testing in clinical trials — http://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2020_09_HMA_CTFG_Contraception_guidance_Version_1.1_updated.pdf
- See also: European Medicines Agency Assessment Report for Paxlovid — http://www.ema.europa.eu/en/documents/assessment-report/paxlovid-epar-public-assessment-report_en.pdf
- See also: Information related to Paxlovid — http://www.pfizer.com
- See also: Late breaking abstract 2021 ERS International Congress - Early follow-up of hospitalised and non-hospitalised patients with Covid-19 in a Swedish setting — http://erj.ersjournals.com/content/58/suppl_65/PA487